CLINICAL TRIAL: NCT04672382
Title: Effect of Intradermal Morphine Application on Histaminergic and Non-histaminergic Itch and Related TRPV1 and Antihistamine Treatment
Brief Title: Evaluation of Peripheral Itch Mechanisms Following Injection of Morphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, PhD, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20200084
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Morphine; Histamine; Cowhage; Isotonic Saline
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morphine (Experimental): During the 1st session, each of the middle forearms of the subject will be divided into two squared areas (4x4 cm) located 3 cm apart. Two areas will be treated with an intradermal injection of morphine (0.05 ml, 0.1 mg/ml), while two areas will be treated with injections of isotonic saline (0.05 ml, 0.9%) as vehicle. Fifteen minutes after the injections, the measurement of FLPI and wheal size will be conducted in one morphine and one saline treated area.
  This measurement will be followed by application of histamine and cowhage in the four areas (two pre-treated with morphine and two pre-treated with vehicle)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — During the 1st session, each of the middle forearms of the subject will be divided into two squared areas (4x4 cm) located 3 cm apart. Two areas will be treated with an intradermal injection of morphine (0.05 ml, 0.1 mg/ml), and two areas with an intradermal injection of isotonic saline.

SUMMARY:
The aim of this study is to the effect of opioid (morphine) intradermal application on histaminergic and non-histaminergic itch. In particular, we would like to demonstrate that also peripheral administration of morphine may affect mast cell release of histamine.

DETAILED DESCRIPTION:
Opioids (i.e. substances extracted from opium poppies, e.g. morphine) are used for treatment of both acute and chronic pain conditions as well as in surgical procedures. Opioids render effective pain relief, however, they may cause bothersome itch as a side effect. With this series of experiments, we wish to clarify how an injection with morphine in the skin layer called dermis (located right below the upper skin) will affect itch.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Participants with any clinically significant abnormalities that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other addictive drugs
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics and pain killers as well as systemic or topical steroids.
* Participants with known allergy/discomfort to the opioid morphine and antihistamine.
* Skin diseases
* Moles, scars or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring itch by computerized Visual Analog Scale Scoring | 10 minutes
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Measuring pain by computerized Visual Analog Scale Scoring | 10 minutes
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Superficial blood perfusion measurement | 15 minutes
  Superficial blood perfusion is measured by a Speckle contrast imager

SECONDARY OUTCOMES:
While size | 15 minutes
  While size will be assessed with a ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Lo Vecchio, Aalborg, North Denmark, Denmark